CLINICAL TRIAL: NCT01946906
Title: Effects of Rifaximin, by Modulation of the Gut Microbiota, on Markers of Systemic Inflammation in Patients With Common Variable Immunodeficiency - An Exploratory Open-label Randomized Controlled Trial
Brief Title: The Rifaximin Study in CVID
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Børre Fevang, Dr, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2013/1037; 2013-000883-27 (EudraCT Number); 13/09446-7 (Other: The Norwegian Medicines Agency)
Record Dates: First submitted 2013-09-12; First posted 2013-09-20 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2014-11

CONDITIONS: Common Variable Immunodeficiency (CVID)
MeSH Terms: conditions — Common Variable Immunodeficiency | interventions — Rifaximin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- No treatment (No Intervention): patient receive no active treatment
- Rifaximin (Experimental): Patient takes Rifaximin 550mg twice daily for 14 days
  Interventions: Drug: Rifaximin

INTERVENTIONS:
Drug: Rifaximin
  Other Names: Xifaxan
  Arms: Rifaximin

SUMMARY:
Patients with Common variable immunodeficiency (CVID) have various forms of autoimmune and auto inflammatory disorders. The study will investigate if intervention with Rifaximin modifies the gut microbiota with a subsequent alteration in markers of systemic immune activation and inflammation in patients with CVID. The investigators hypothesize that the gut microbiota of CVID patients, at least partly through interaction with the innate immune system within the intestine, contribute to a low-grade systemic inflammation in these patients, and that an intervention with the non-absorbable antibiotic Rifaximin attenuates systemic inflammation through modulation of the gut microbiota. The study may lead to increased understanding of the interaction between microbiota and the immune system. The study could give new insight into important disease processes in relation to the interaction between the microbiota, the intestine and the systemic compartment, and potentially be the basis of new therapeutic strategies in these patients to prevent and down-regulate the auto-inflammatory and autoimmune complications seen in CVID. The findings could also be of relevance for other disorders where the interaction between microbiota and intestinal and systemic inflammation is involved such as various cardiovascular and metabolic disorders.

The investigators hypothesize that the gut microbiota of CVID patients, at least partly through interaction with the innate immune system within the intestine, contribute to a low-grade systemic inflammation in these patients, and that an intervention with the non-absorbable antibiotic Rifaximin attenuates systemic inflammation through modulation of the gut microbiota.

ELIGIBILITY:
Inclusion Criteria:

* 18 ≥ and <75 years of age
* A diagnosis of CVID: decreased serum levels (> 2 SD) of immunoglobulin (Ig)G, IgA and/or IgM and exclusion of other forms of hypogammaglobulinemia

Exclusion Criteria:

* Previous treatment with antibiotics within the last 12 weeks
* History of hypersensitivity to Rifaximin or other Rifamycin derived antimicrobial agents, or any of the components of XIFAXAN
* Comorbidity not related to CVID- i.e. conditions or symptoms that may influence with the patient safety or compromise the study results (e.g., cardiovascular disorders, alcoholism, psychiatric disease, HIV infection etc.)].
* Polypharmacy with increased risk for interactions. i.e. patient with an extensive medication lists (e.g. 10 drugs or more) this may influence with the patient safety or compromise the study results
* Malignancy of any cause
* Impaired kidney function (i.e., estimated glomerulus filtration rate <50 ml/minute/1.73 m2]
* Impaired liver function (Alanine aminotransferase > 150 U/l) or established liver cirrhosis.
* Pregnant or planning to be pregnant in the study period to avoid interference of pregnancy with gut microbiota (not because of toxicity].
* Nursing
* On-going infection, including GI infection
* The use of probiotics for the recent 6 months
* Any immunosuppressive drugs,

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Changes in inflammatory and anti-inflammatory mediators | after 2 and 8 weeks after Day 0
  Changes in serum/plasma/whole blood of tumor necrosis factor alpha (TNF-alpha), c reactive protein (CRP), soluble CD14 and other cytokines/chemokines.

CONTACTS AND LOCATIONS:
Overall Officials: Borre Fevang, MD, Phd, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway